CLINICAL TRIAL: NCT04764305
Title: Liver Disease, Myocardial Fibrosis and Collaterals in the Adult Fontan Patient - a Metabolomics and Proteomics Approach
Brief Title: Liver Disease, Myocardial Fibrosis and Collaterals in the Adult Fontan Patient a Metabolomics and Proteomics Approach
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other); Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, OÄ Dr. Miriam Michel, Principal Investigator, Medical University Innsbruck
Other Study IDs: registration in progress
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Patient Participation; Heart Defects, Congenital; Liver Diseases; Collateral Circulation, Any Site; Myocardial Fibrosis
Keywords: Fontan; congenital heart disease; inflammation; Fontan-associated liver disease; Myocardial fibrosis; Collateral vessel
MeSH Terms: conditions — Patient Participation; Heart Defects, Congenital; Liver Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with Fontan circulation. No intervention planned (observational study)
- Controls: Healthy, biventricular controls. No intervention planned (observational study)

SUMMARY:
Out objective is to identify the mechanisms that promote hepatic and myocardial fibrosis, and collateral vessel formation in patients with complex congenital heart disease and Fontan circulation.

DETAILED DESCRIPTION:
In their prior works the investigators could show that there is evidence of a proinflammatory condition in a certain subgroup of patients with complex congenital heart disease and a so called Fontan circulation. Those patients are also prone to develop hepatic and myocardial fibrosis as well as to reveal collateral vessel formation. The investigators' hypothesis is that this pro-inflammatory condition is not only reflecting pre-stages of one or more of those 3 issues, but that this is also a main driving mechanism to develop and hepatic or myocardial fibrosis and collateral vessels.

The objective of the here proposed study thus is to identify the mechanisms that promote hepatic and myocardial fibrosis, and collateral vessel formation, and thus provide insight into the determination of those Fontan patients that tend to develop those conditions. The investigators attempt to link the issues of hepatic and myocardial fibrosis and collateral vessel formation by directing our focus on the phospholipid, amino acid and bile acid metabolism and on cell surface markers, cytokines, and chemokines as surrogates for proinflammatory, profibrotic and proangiogenic conditions.

This study would thereby allow for a deeper insight into Fontan pathophysiology and sequelae and might provide first steps towards the identification of possible diagnostic or eventually therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent of participants
* age at testing of ≥18 years
* 8 h fasting before blood sampling
* Fontan circulation (patients)
* biventricular heart without structural or functional abnormality (controls)

Exclusion Criteria:

* Protein losing enteropathy (PLE) (patients are defined as "PLE positive" if there is/are serum protein <5g/dL and serum albumin <3g/dL (duration for more than 3 months and exclusion of other causes for hypoproteinemia) and documented enteric protein loss: faecal alpha-1-antitrypsin ≥400 µg/g
* medication directly affecting metabolic state, such as cholesterol-lowering agents, or haemodynamic state, such as beta-blockers or sildenafil, with the exception of angiotensin converting enzyme inhibitors, diuretics, and anticoagulants
* atrial or ventricular arrhythmia
* coronary artery disease (history of myocardial infarction, myocardial revascularisation, percutaneous coronary intervention, or coronary artery bypass surgery)
* any metabolic disease, such as diabetes mellitus
* malignancy
* obesity (body mass index (BMI) >25 kg/m2)
* underweight (BMI < 18 kg/m2)
* renal disease
* inflammatory disease such as acute or chronic infection
* myeloproliferative disorder
* pregnancy or lactation
* malnourishment
* mental handicap not allowing valid consent to participation in the study or CMR
* need of sedation or general anesthesia for CMR
* typical contraindications for performing CMR such as metal-containing mechanical or electronic implants
* claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with Fontan circulation, see inclusion criteria. Healthy, biventrucal age- and sex-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants | July 2021-December 2023
  When aspired number of participants is reached

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Michel, MD, Principal Investigator — Medical University of Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No